CLINICAL TRIAL: NCT04804384
Title: Assessment of the Functional Impact of a Closed-loop Controlled Prehension Neuroprosthesis in Post-stroke Patients. PREHENS-STROKE
Brief Title: Assessment of the Functional Impact of a Close-loop Controlled Prehension Neuroprosthesis in Post-stroke Patients
Acronym: PREHENS-STROKE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: RC31/19/0502
Record Dates: First submitted 2021-03-09; First posted 2021-03-18 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental (Experimental)
  Interventions: Device: Prehension neuroprosthesis

INTERVENTIONS:
Device: Prehension neuroprosthesis — The experimental condition corresponds to patients in the condition where the prehension neuroprosthesis is active, which means that the extensor muscles of the fingers and thumb will be stimulated by the prehension neuroprosthesis to ensure the opening of the hand. The prehension neuroprosthesis designates a functional electrical stimulation device controlled by the patient which will itself trigger the stimulation of the extensor muscles of the fingers (closed-loop control), according to stimuli which it controls voluntarily. The goal is to restore an opening of the fingers to capture objects.
  The control condition corresponds to the patients in the condition where the prehension neuroprosthesis is inactive.

SUMMARY:
The aim of the PREHENS-STROKE study is to propose a functional replacement device to restore grip capacities in patients with hemiparesis after stroke, unable to actively open the hand to seize objects. The main objective is to evaluate the impact of the use of a self-controlled prehension neuroprosthesis on the ability to perform a standardized grasping task, consisting of grasping, relocating and releasing a glass (palmar grasp) or a spoon (key-pinch), compared to a condition without the use of the prehension neuroprosthesis.

DETAILED DESCRIPTION:
Stroke is the leading cause of motor impairment acquired after 40 years. Of the affected patients, 50% do not recover active finger extension and there is no satisfactory solution for functional recovery of the grip in these patients. The use of wearable exoskeletons to improve the grip is limited by their size and cost. An alternative is the use of functional electrical stimulation of the grasping muscles, named prehension neuroprosthesis, well developed in the spinal cord injured patient. In the adult hemiplegic patient, only about ten studies concerned the functional impact of a prehension neuroprosthesis, which have shown potential to perform a correct hand opening linked with a significant functional gain. Nevertheless, one of the major problems concerns the definition of the optimal modalities to control the prehension neuroprosthesis, modalities which until now have proved unsuitable for post-stroke patients: an open-loop control with manual triggering of the neuroprosthesis (press-button type) is not suitable with daily living use; control with the contralateral upper-limb is also not suitable for everyday use where bimanual tasks are required; and finally, the use of the residual voluntary electromyographic activity of the targeted muscle limits the opening of the fingers and the reliability of the control by promoting the occurrence of spastic cocontractions of the flexors of the fingers.

In this context, the present project proposes to evaluate the functional contribution of a closed-loop controlled prehension neuroprosthesis that will restore an extension of the fingers and the thumb in order to improve the grip function.

Each patient is evaluated 5 times during visits lasting between 1h30 and 2 hours. Patients are already admitted to standard care for a period of at least 5 consecutive days in the Rehabilitation Center. The visit (Day 1) will include the patient and collect the Action Arm Research Test (ARAT) and Upper Limb Performance Assessment (ULPA) scores achieved with the inactive prehension neuroprosthesis. The visit T1 (day 2) will select the preferred control mode of the neuroprosthesis. The visit T2 (day 3) and T3 (day 4) will allow learning and training in the use of the neuroprosthesis. The visit T4 (day 5) will evaluate the functional impact of the neuroprosthesis: the patients will perform the standardized primary and secondary gripping tasks with the activated or inactivated neuroprosthesis, then the ARAT and ULPA with activated neuroprosthesis, and finally the Psychosocial Impact of Assistive Devices Scale and the Device subscale of the Quebec User Assessment of Satisfaction with Assistive Technology questionnaire will be completed. The end of the visit T4 corresponds to the end of the patient's inclusion in the research protocol.

ELIGIBILITY:
Inclusion Criteria:

* Concerning the study population: Paresis of an upper limb from a single ischemic or hemorrhagic, hemispheric or brainstem stroke, as evidenced by brain imaging (CT or MRI); Stroke more than one month old; Impossibility to actively expand the fingers 2 to 5 (opening of the hand) to intentionally grab an empty glass (identical to the material used for the Action Research scale Arm Test), with a palmar grip (cylindrical grip), while the subject can hold the glass passively placed in the hand and/or the thumb to voluntarily grab the handle of a tablespoon (flat, like a wrench) with a key-grip (identical to that of the Wolf Motor Function Test), while the subject can hold the spoon previously placed passively between thumb and index; Ability to sit on a chair at least during 1h30.
* Concerning legislative aspects: Free, informed and written consent signed by the participant and the investigator (at the latest on the day of inclusion and before any investigation required by the research); Affiliate or beneficiary of the French health insurance system; The person is of age (at least 18 years old); Women and men are included; The patient is available for a follow-up of 5 days as part of his hospitalization performed as part of routine care.

Exclusion Criteria:

* Concerning the study population: The person is parturient, or is breastfeeding; The person is pregnant, the diagnosis being guided by the interrogation (date of the last menstruation, desire of pregnancy, contraception) and possibly confirmed by a blood test (beta hCG); Musculotendinous retractions or joint stiffness of the fingers and wrist preventing passive opening of the hand sufficient to perform at least one of the functional tasks evaluated; Limitation of the approach which does not make it possible to carry out the task of gripping in front of the trunk, the subject sitting; Upper limb pain limiting achievement of the primary standardized grasping task; Major sensory disorders corresponding to a sub-score Somesthesia of the modified Erasmus Nottingham Sensory Assessment French version (EmNSA-F) for the upper limb <10/44; Severe aphasia with aphasia severity scale of the Boston Diagnostic Severity Aphasia Examination, indicating that there may be a clear decrease in verbal fluency or ease and speed of understanding, with no significant limitation expression or communication; Unilateral spatial negligence highlighted with the bells test if the difference between the omissions in the left and right fields is greater than or equal to 6; Extensor digitorum communis muscle and/or pollicis extensor longus muscle not stimulable with the neuroprosthesis, i.e. a sufficient extension of fingers and/or thumb for grasping tasks is not obtained with an electrical stimulation well supported by the patient.
* Concerning the associated pathologies: The person is carrying a pacemaker; Presence of unstable epilepsy; Presence of unstable cardio-vascular disease (coronary heart disease, major hypertension, heart failure); Presence of a dermatological problem against indicating the application of surface electrodes.
* Concerning associated treatments: The person should not receive an injection of botulinum toxin in the upper limb during the period of inclusion in the protocol, or in the 30 days prior to inclusion.
* Concerning legislative aspects: The person is participating in another research protocol including an exclusion period still in progress; The person is under the protection of justice or guardianship; The person refuses to sign the consent; It is not possible to give the person informed information and to make sure of the subject's compliance due to impaired physical and/or psychological health.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-08-30 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Success rate of a main standardized gripping task performed | 5 days
  The primary endpoint is a comparison of the success rate of a main standardized gripping task performed with the activated and inactivated prehension neuroprosthesis. This task consists of grasping, moving and releasing either an object with a palmar grasp (glass) or a key grip between thumb and index (to catch the handle of a spoon or a key). During the visit T3, the patient chooses the main functional task from the two standardized tasks (the other becomes the secondary task). The evaluation consists of 24 trials with active or inactive prehension neuroprosthesis (12 activated and 12 inactivated). The criterion selected as a success corresponds to the success of at least 70 percent of the tests, i.e. 8 out of 12 trials in each condition. This success / failure score is made from video recordings, by an evaluator blinded to the activation or not of the prehension neuroprosthesis, from data collected during the visit T4 (5th and last day).

SECONDARY OUTCOMES:
Comparison of success rate | 5 days
  Comparison of success rate when performing the secondary standardized gripping task performed with the activated and inactivated prehension neuroprosthesis. Evaluation is identical to the main standardized gripping task. This success / failure score is made from video recordings, by an evaluator blinded to the activation or not of the prehension neuroprosthesis, from data collected during the visit T4 (5th and last day).
Qualitative analysis | 2 days
  Qualitative analysis of the reasons for choosing the prehension neuroprosthesis closed-loop control modalities, among the 6 modalities initially proposed, carried out during the visit T1 (second day).
Analysis of the quality | 5 days
  Analysis of the quality (rated between 0 and 5) of the capture, transport and release phases, during each test of the main and secondary standardized gripping tasks (data collected during visit T4). The assessment is made in a delayed manner from video recordings, by an evaluator blinded to the activation or not of the prehension neuroprosthesis. An analysis according to the n-of-1 trials methodology is performed to determine the link between activation / inactivation of the prehension neuroprosthesis and the quality and duration of the movement studied.
Analysis of the the duration | 5 days
  Analysis of the the duration (in seconds) of the capture, transport and release phases, during each test of the main and secondary standardized gripping tasks (data collected during visit T4). The assessment is made in a delayed manner from video recordings, by an evaluator blinded to the activation or not of the prehension neuroprosthesis. An analysis according to the n-of-1 trials methodology is performed to determine the link between activation / inactivation of the prehension neuroprosthesis and the quality and duration of the movement studied.
Comparison of the Action Research Arm Test score | 5 days
  Comparison of the Action Research Arm Test score (ARAT, score between 0 and 57, evaluation of different unimanual grip modes) performed with the inactivated (visit T0) and activated (visit T4) prehension neuroprosthesis. The assessment is made in a delayed manner from video recordings, by an evaluator blinded to the activation or not of the prehension neuroprosthesis.
Comparison of the Upper Limb Performance Assessment score | 5 days
  Comparison of the Upper Limb Performance Assessment score (ULPA, score 0 to 100, evaluation of bimanual hand grips) performed with the inactivated (visit T0) and activated (visit T4) prehension neuroprosthesis. The assessment is made in a delayed manner from video recordings, by an evaluator blinded to the activation or not of the prehension neuroprosthesis.
Evaluation of the effect of the prehension neuroprosthesis | 5 days
  Evaluation of the effect of the prehension neuroprosthesis in the person's life with the 3 subscales (competence, adaptability and self-esteem) of the score Psychosocial Impact of Assistive Devices Scale (F-PIADS, score between - 3 and +3 for each subscale). Data collected during the visit T4.
Evaluation of the patient satisfaction and tolerance | 5 days
  Evaluation of the patient satisfaction and tolerance to the use of the prehension neuroprosthesis with the Device subscale of the Quebec User Assessment of Satisfaction with Assistive Technology (QUEST, scoring between 0 and 5). Data collected during the visit T4.
Evaluate the modification of the brain activations | 5 days
  Evaluate the modification of the brain activations (localization of maximum desynchronization) recorded by electroencephalography, during the performance of a standardized functional task (similar to the main a standardized functional task) with and without NAP. Data collected during the visit T4.

CONTACTS AND LOCATIONS:
Overall Officials: David GASQ, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital, Toulouse, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Le Guillou R, Froger J, Morin M, Couderc M, Cormier C, Azevedo-Coste C, Gasq D. Specifications and functional impact of a self-triggered grasp neuroprosthesis developed to restore prehension in hemiparetic post-stroke subjects. Biomed Eng Online. 2024 Dec 21;23(1):129. doi: 10.1186/s12938-024-01323-y. PMID 39709421